CLINICAL TRIAL: NCT01888978
Title: A Pilot Study of Molecularly Tailored Therapy for Patients With Metastatic Pancreatic Cancer
Brief Title: Molecularly Tailored Therapy for Pancreas Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-384
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2017-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas; cancer; metastatic; chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine; Oxaliplatin; Fluorouracil; Docetaxel; Leucovorin; IFL protocol; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Modified FOLFOX-6 (Experimental): Oxaliplatin 85 mg/m2 day 1 and 5-fluorouracil 400 mg/m2 day 1 and Leucovorin 400 mg/m2 day 1 and 5-fluorouracil 2400 mg/m2 over 46 hours on day 1-3 of every 14 day cycle All drugs will be administered until disease progression or unacceptable toxicity are observed
  Interventions: Drug: Modified FOLFOX-6
- Ox-Tax (Experimental): Docetaxel 65 mg/m2 and Oxaliplatin 100 mg/m2 on day 1 every 3 weeks All drugs will be administered until disease progression or unacceptable toxicity are observed
  Interventions: Drug: Ox-Tax
- FOLFIRI (Experimental): Irinotecan 180 mg/m2 on day 1 and 5-FU 400 mg/m2 on day 1 and Leucovorin 400 mg/m2 day 1 and 5-FU 2400 mg/m2 over 46 hours, days 1-3 as a continuous infusion All drugs will be administered until disease progression or unacceptable toxicity are observed
  Interventions: Drug: FOLFIRI
- Tax-Iri (Experimental): 2 weeks on, 1 week off of Docetaxel 35 mg/m2/week and Irinotecan 50 mg/m2/week Both administered on day 1 of each week of treatment All drugs will be administered until disease progression or unacceptable toxicity are observed
  Interventions: Drug: Tax-Iri
- Gem-Ox (Experimental): Gemcitabine: 1000 mg/m2 over 100 minutes on Day 1 Oxaliplatin: 100 mg/m2 over 120 minutes on Day 2 of every 14 day cycle All drugs will be administered until disease progression or unacceptable toxicity are observed
  Interventions: Drug: Gem-OX
- Gem-5FU (Experimental): Gemcitabine: 1000 mg/m2 over 30 minutes 5-FU 2000/m6 as a 24 hour infusion on days 1, 8, and 15 of every 28 day cycle All drugs will be administered until disease progression or unacceptable toxicity are observed
  Interventions: Drug: Gem-5FU
- Gem-Tax (Experimental): Gemcitabine 1000 mg/m2 over 30 minutes and Docetaxel 35 mg/m2 over 60 minutes on days 1, 8, and 15 of every 28 day cycle
  Interventions: Drug: Gem-Tax

INTERVENTIONS:
Drug: Gem-OX
  Other Names: Gemcitabine; Gemzar; Oxaliplatin; Eloxatin
  Arms: Gem-Ox
Drug: Gem-5FU
  Other Names: Gemcitabine; Gemzar; 5-FU; 5-fluorouracil
  Arms: Gem-5FU
Drug: Gem-Tax
  Other Names: Gemcitabine; Gemzar; Docetael; taxotere
  Arms: Gem-Tax
Drug: Modified FOLFOX-6
  Other Names: Oxaliplatin; Eloxatin; 5-FU; 5-Fluorourcil; Leucovorin
  Arms: Modified FOLFOX-6
Drug: Ox-Tax
  Other Names: Docetaxel; Taxotere; Oxalipaltin; Eloxatin
  Arms: Ox-Tax
Drug: FOLFIRI
  Other Names: Irinotecan; CPT-11; 5-FU; 5-Fluorouracil; Leucovorin
  Arms: FOLFIRI
Drug: Tax-Iri
  Other Names: Docetaxel; Taxotere; Irinotecan; CPT-11
  Arms: Tax-Iri

SUMMARY:
Patient therapy is tailored according to the molecular profile of the patient's tumor.

DETAILED DESCRIPTION:
This study is for patients with metastatic pancreatic cancer (cancer that has spread to other parts of the body). The purpose of this study is to determine whether molecularly tailored therapy can improve the effectiveness of standard chemotherapy combinations for patients with metastatic pancreatic cancer. A series of special tests will be performed on a sample of tumor, and based on the results subjects will be assigned to one of seven chemotherapy treatments, with each being the combination of two standard chemotherapies. Each of these combinations has been safely used in patients with pancreatic or other types of cancer. The purpose of this study is to to determine the ability to personalize therapy in this manner, and to determine how many patients a larger study would need. A second purpose is not to determine if one doublet is better than another. Rather, this second purpose is to show that for all patients enrolled in this protocol who have been assigned a doublet based on their tumor's molecular analysis (molecular tailoring), treatment response will be better than would be expected compared to patients who have been treated in the past with no molecular tailoring.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven pancreatic adenocarcinoma with measurable disease
* Biopsy accessible tumor deposits
* ECOG performance status 0-2
* Age >/= 18 years
* Subjects with no brain metastases or history of previously treated brain metastases
* Adequate hepatic, renal, and bone marrow function
* Partial thromboplastin time must be </= 1.5 x upper normal limit of institution's normal range and INR < 1.5
* Life expectancy > 12 weeks
* Women of childbearing potential must have a negative seum pregnancy test within 14 days prior to initiation of treatment
* Subject is capable of understanding and complying with parameters as outlines in the protocol and able to sign and date the consents

Exclusion Criteria:

* CNS metastases which do not meet criteria outlines in inclusion criteria
* Active severe infection or known chronic infection with HIV or hepatitis B virus
* Cardiovascular disease
* Life threatening visceral disease or other severe concurrent disease
* Women who are pregnant, breastfeeding, or women of childbearing potential not using dual forms of effective contraception
* Anticipated patient survival under 3 months
* Patients receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biological composition to gemcitabine, oxaliplatin, 5-FU, docetaxel or irinotecan
* Uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-12; Primary Completion 2016-06 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Timing of biopsy and treatment | 1 year
  The number of days from study entry to biopsy to molecular results to first dose

SECONDARY OUTCOMES:
Estimates for future trials | 1 year
  objective response rate, proportions of patients with each molecular profile, timing of biopsy and therapy results, usefulness of molecular profile results and adverse events.
Clinical Benefit | 1 year
  confirmed classification of stable disease, partial response, or complete response
Progression-free survival | 1 year
  Time in days from study entry until progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pishvaian, MD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Georgetown University- Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - MedStar Montgomery Medical Center, Olney, Maryland